CLINICAL TRIAL: NCT02912260
Title: A Phase 2, Multi-Center, Double-Blind, Randomized, Placebo-controlled Study of MGL-3196 in Patients With Non-alcoholic Steatohepatitis
Brief Title: Phase 2 Study of MGL-3196 in Patients With Non-Alcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Madrigal Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MGL-3196-05
Record Dates: First submitted 2016-09-19; First posted 2016-09-23 (Estimated); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-09

CONDITIONS: Non-alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — resmetirom

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MGL-3196 (Experimental): Study Drug
  Interventions: Drug: MGL-3196
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MGL-3196
  Arms: MGL-3196
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine the effect of once-daily oral MGL-3196 on the percent change in hepatic fat fraction from baseline in participants with biopsy-proven Non-alcoholic Steatohepatitis (NASH).

ELIGIBILITY:
Inclusion Criteria. Participants who meet all of the following criteria will be eligible to participate in the study:

* Must be willing to participate in the study and provide written informed consent;
* Male and female adults ≥18 years of age;
* Female participants of child bearing potential with negative serum pregnancy (beta human chorionic gonadotropin) tests who are not breastfeeding, do not plan to become pregnant during the study, and agree to use effective birth control (that is, condoms, diaphragm, nonhormonal intrauterine device [IUD], or sexual abstinence [only if this is in line with the participant's current lifestyle]) throughout the study and for at least 1 month after study completion; hormonal contraception (estrogens stable ≥3 months) and hormonal IUDs are permitted if used with a secondary birth control measure (for example, condoms); or female participants of non-child bearing potential (that is, surgically [bilateral oophorectomy, hysterectomy, or tubal ligation] or naturally sterile [>12 consecutive months without menses]); Male participants who have sexual intercourse with a female partner of child bearing potential from the first dose of study drug until 1 month after study completion must be either surgically sterile (confirmed by documented azoospermia >90 days after the procedure) or agree to use a condom with spermicide. All male participants must agree not to donate sperm from the first dose of study drug until 1 month after study completion;
* Must have confirmation of ≥10% liver fat content on magnetic resonance imaging proton density fat fraction;
* Biopsy-proven NASH. Must have had prior liver biopsy within 180 days of randomization with fibrosis stage 1 to 3 and a non-alcoholic fatty liver disease activity score (NAS) of ≥4 with a score of 1 or more in each of the following NAS components:

  * Steatosis (scored 0 to 3),
  * Ballooning degeneration (scored 0 to 2), and
  * Lobular inflammation (scored 0 to 3);
* Must have documented historical (3 weeks to 6 months prior to the study entry) alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels consistent with the screening ALT and AST values.

Exclusion Criteria. Participants who meet any of the following criteria will be excluded from participation in the study:

Note: Unless otherwise specified, repeat testing may be performed in consultation with the Medical Monitor.

* History of significant alcohol consumption for a period of more than 3 consecutive months within 1 year prior to screening;
* Hyperthyroidism;
* Participants on thyroid replacement therapy (with exceptions);
* Prior or planned (during the study period) bariatric surgery (for example, gastroplasty, roux-en-Y gastric bypass);
* Type 1 diabetes;
* Uncontrolled Type 2 diabetes defined as Hemoglobin A1c (HbA1c) ≥ 9.5% at screening (participants with HbA1c ≥ 9.5% may be rescreened);
* Use of obeticholic acid, ursodeoxycholic acid (Ursodiol® and Urso®), high dose vitamin E (>400 IU/day) unless on stable dose of vitamin E >400 IU/day for at least 6 months at the time of liver biopsy, or pioglitazone within 90 days prior to enrollment or since screening biopsy, whichever is longer;
* Presence of cirrhosis on liver biopsy (stage 4 fibrosis);
* Platelet count < 140,000/mm^3;
* Clinical evidence of hepatic decompensation;
* Evidence of other forms of chronic liver disease;
* Active, serious medical disease with likely life expectancy <2 years;
* Participation in an investigational new drug trial in the 30 days prior to randomization; or
* Any other condition which, in the opinion of the Investigator, would impede compliance, hinder completion of the study, compromise the well-being of the participant, or interfere with the study outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2016-10-18 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2021-11-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Madrigal Research Site, Dothan, Alabama
  - Madrigal Research Site, Tucson, Arizona
  - Madrigal Research Site, Coronado, California
  - Madrigal Research Site, Los Angeles, California
  - Madrigal Research Site, Rialto, California
  - Madrigal Research Site, San Diego, California
  - Madrigal Research Site, Ventura, California
  - Madrigal Research Site, Englewood, Colorado
  - Madrigal Research Site, Boca Raton, Florida
  - Madrigal Research Site, Lakewood Rch, Florida
  - Madrigal Research Site, Lauderdale Lakes, Florida
  - Madrigal Research Site, Miami, Florida
  - Madrigal Research Site, New Port Richey, Florida
  - Madrigal Research Site, Kansas City, Kansas
  - Madrigal Research Site, Monroe, Louisiana
  - Madrigal Research Site, Baltimore, Maryland
  - Madrigal Research Site, Jackson, Mississippi
  - Madrigal Research Site, St Louis, Missouri
  - Madrigal Research Site, Albuquerque, New Mexico
  - Madrigal Research Site, New York, New York
  - Madrigal Research Site, Durham, North Carolina
  - Madrigal Research Site, Rapid City, South Dakota
  - Madrigal Research Site, Live Oak, Texas
  - Madrigal Research Site, San Antonio, Texas
  - Madrigal Research Site, Charlottesville, Virginia
  - Madrigal Research Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harrison SA, Ratziu V, Anstee QM, Noureddin M, Sanyal AJ, Schattenberg JM, Bedossa P, Bashir MR, Schneider D, Taub R, Bansal M, Kowdley KV, Younossi ZM, Loomba R. Design of the phase 3 MAESTRO clinical program to evaluate resmetirom for the treatment of nonalcoholic steatohepatitis. Aliment Pharmacol Ther. 2024 Jan;59(1):51-63. doi: 10.1111/apt.17734. Epub 2023 Oct 2. PMID 37786277
- [Derived] Younossi ZM, Stepanova M, Taub RA, Barbone JM, Harrison SA. Hepatic Fat Reduction Due to Resmetirom in Patients With Nonalcoholic Steatohepatitis Is Associated With Improvement of Quality of Life. Clin Gastroenterol Hepatol. 2022 Jun;20(6):1354-1361.e7. doi: 10.1016/j.cgh.2021.07.039. Epub 2021 Jul 27. PMID 34329774
- [Derived] Harrison SA, Bashir M, Moussa SE, McCarty K, Pablo Frias J, Taub R, Alkhouri N. Effects of Resmetirom on Noninvasive Endpoints in a 36-Week Phase 2 Active Treatment Extension Study in Patients With NASH. Hepatol Commun. 2021 Jan 4;5(4):573-588. doi: 10.1002/hep4.1657. eCollection 2021 Apr. PMID 33860116
- [Derived] Harrison SA, Bashir MR, Guy CD, Zhou R, Moylan CA, Frias JP, Alkhouri N, Bansal MB, Baum S, Neuschwander-Tetri BA, Taub R, Moussa SE. Resmetirom (MGL-3196) for the treatment of non-alcoholic steatohepatitis: a multicentre, randomised, double-blind, placebo-controlled, phase 2 trial. Lancet. 2019 Nov 30;394(10213):2012-2024. doi: 10.1016/S0140-6736(19)32517-6. Epub 2019 Nov 11. PMID 31727409

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants underwent screening procedures within 42 days of randomization. To participate in the study, participants were required to have had a qualifying liver biopsy within 180 days of randomization.
Groups:
- MGL-3196: Randomized participants received MGL-3196 80 mg orally once daily in the morning for 36 weeks.
- Placebo: Randomized participants received matching placebo orally once daily in the morning for 36 weeks.
Period: Main Study
Arm/Group | MGL-3196 | Placebo
Started | 84 | 41
Received at Least 1 Dose of Study Drug | 84 | 41
Completed | 74 | 34
Not Completed | 10 | 7
Not completed — Lost to Follow-up | 5 | 4
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Adverse Event | 3 | 0
Not completed — Physician Decision | 0 | 1
Period: Extension Study
Arm/Group | MGL-3196 | Placebo
Started | 17 | 14
Completed | 16 | 13
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MGL-3196 | Placebo | Total
Number analyzed (Participants) | 84 | 41 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (10.35) | 47.3 (11.71) | 50.3 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 17 | 63
  Male | 38 | 24 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 22 | 59
  Not Hispanic or Latino | 47 | 19 | 66
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 80 | 37 | 117
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Hepatic Fat Fraction by MRI-PDFF at Screening [Mean (Standard Deviation); unit: percentage] | 20.25 (6.843) | 19.63 (8.159) | 20.05 (7.274)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline To Week 12 In Hepatic Fat Fraction Assessed By Magnetic Resonance Imaging Proton Density Fat Fraction (MRI-PDFF)
Description: The primary endpoint was relative change in MRI-PDFF assessed hepatic fat fraction compared with placebo at Week 12 in participants who had both a baseline and Week 12 MRI-PDFF. Least squares (LS) mean was provided for the statistical comparison of MGL-3196 versus placebo.
Time Frame: Week 12
Population: MRI-PDFF evaluable population: all participants who were randomized in the study, received study drug, and finished Week 12 visit, with valid MRI-PDFF measurements at both baseline and Week 12 Visit.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 78 | 38
percent change | -32.9 (3.0) | -10.4 (4.3)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; LS mean difference in hepatic fat fraction between MGL-3196 and placebo at Week 12; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Net) = -22.5, 95% CI 2-sided [-32.9 to -12.2], Standard Error of Mean 5.22

2. Secondary Outcome: Percentage Of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, which does not necessarily have a causal relationship with the treatment. A summary of serious and all other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Week 12 and Week 36
Population: Safety population: all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 84 | 41
percentage of participants
  Week 12 | 71.4 | 46.3
  Week 36 | 86.9 | 68.3

3. Secondary Outcome: Percent Change From Baseline To Week 36 In Hepatic Fat Fraction Assessed By MRI-PDFF
Description: The endpoint was relative change assessed hepatic fat fraction compared with placebo at Week 36. LS mean was provided for the statistical comparison of MGL-3196 versus placebo.
Time Frame: Week 36
Population: Modified Intent-to-Treat (mITT) population: all participants who were randomized in the study, received at least 1 dose of study drug, and had lipid and other efficacy measurements at Week 4 or later visits.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 74 | 34
percent change | -37.3 (3.7) | -8.9 (5.4)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; LS mean difference in hepatic fat fraction between MGL-3196 and placebo at Week 36; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Net) = -28.4, 95% CI 2-sided [-41.3 to -15.4], Standard Error of Mean 6.52

4. Secondary Outcome: Change From Baseline To Week 12 In Absolute Hepatic Fat Fraction Assessed By MRI-PDFF
Description: The endpoint was change in MRI-PDFF assessed absolute hepatic fat fraction compared with placebo at Week 12. LS mean was provided for the comparison of MGL-3196 versus placebo.
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 78 | 38
percentage | -7.0 (0.6) | -2.7 (0.8)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; LS mean difference in absolute hepatic fat fraction between MGL-3196 and placebo at Week 12; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Net) = -4.3, 95% CI 2-sided [-6.3 to -2.4], Standard Error of Mean 0.991

5. Secondary Outcome: Change From Baseline To Week 36 In Absolute Hepatic Fat Fraction Assessed By MRI-PDFF
Description: The endpoint was change in assessed absolute hepatic fat fraction compared with placebo at Week 36. LS mean was provided for the comparison of MGL-3196 versus placebo.
Time Frame: Week 36
Population: mITT population: all participants who were randomized in the study, received at least 1 dose of study drug, and had lipid and other efficacy measurements at Week 4 or later visits.
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 74 | 34
percentage | -8.2 (0.7) | -2.9 (1.0)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; LS mean difference in absolute hepatic fat fraction between MGL-3196 and placebo at Week 36; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Net) = -5.3, 95% CI 2-sided [-7.8 to -2.8], Standard Error of Mean 1.260

6. Secondary Outcome: Percentage Of Participants With At Least 30% Relative Fat Reduction at Week 12
Description: The endpoint presented the percentage of participants achieving a relative fat reduction of ≥30% at Week 12.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 78 | 38
percentage of participants | 60.3 | 18.4

7. Secondary Outcome: Percentage Of Participants With At Least 30% Relative Fat Reduction At Week 36
Description: The endpoint presented the percentage of participants achieving a relative fat reduction of ≥30% at Week 36.
Time Frame: Week 36
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 74 | 34
percentage of participants | 67.6 | 29.4

8. Secondary Outcome: Percentage Of Participants Achieving A 1-Point Reduction In Non-alcoholic Fatty Liver Disease Activity Score (NAS) At Week 36
Description: The NAS is a histologic scale for non-alcoholic steatohepatitis (NASH) activity, which combines into a single score steatosis (Grade 0 to 3), ballooning (Grade 0 to 2), and lobular inflammation (Grade 0 to 3). The endpoint presented the percentage of participants with a 1-point or greater reduction in NAS.
Time Frame: Week 36
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 73 | 34
percentage of participants | 76.7 | 64.7

9. Secondary Outcome: Percentage Of Participants Achieving A 2-Point Reduction In NAS At Week 36
Description: The NAS is a histologic scale for NASH activity, which combines into a single score steatosis (Grade 0 to 3), ballooning (Grade 0 to 2), and lobular inflammation (Grade 0 to 3). The endpoint presented the percentage of participants with a 2-point or greater reduction in NAS.
Time Frame: Week 36
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 73 | 34
percentage of participants | 56.2 | 32.4

10. Secondary Outcome: Percentage Of Participants Achieving A 2-Point Reduction In NAS And Either A ≥1-Point Reduction In Lobular Inflammation Or Hepatocellular Ballooning At Week 36
Description: The NAS is a histologic scale for NASH activity, which combines into a single score steatosis (Grade 0 to 3), ballooning (Grade 0 to 2), and lobular inflammation (Grade 0 to 3). The endpoint presented the percentage of participants with a 2-point or greater reduction in NAS and a 1-point or greater reduction in lobular inflammation or hepatocellular ballooning.
Time Frame: Week 36
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 73 | 34
percentage of participants | 50.7 | 32.4

11. Secondary Outcome: Percentage Of Participants Achieving A 2-Point Reduction In NAS Without Fibrosis Worsening At Week 36
Description: The NAS is a histologic scale for NASH activity, which combines into a single score steatosis (Grade 0 to 3), ballooning (Grade 0 to 2), and lobular inflammation (Grade 0 to 3). Fibrosis stage (0 to 3) was also included in the assessment. The endpoint presented the percentage of participants with a 2-point or greater reduction in NAS without worsening fibrosis.
Time Frame: Week 36
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 73 | 34
percentage of participants | 45.2 | 32.4

12. Secondary Outcome: Percentage Of Participants With A Reduction In Hepatocellular Steatosis At Week 36
Description: The NAS is a histologic scale for NASH activity, which combines into a single score steatosis (Grade 0 to 3), ballooning (Grade 0 to 2), and lobular inflammation (Grade 0 to 3). The endpoint presented the percentage of participants with a reduction in hepatocellular steatosis.
Time Frame: Week 36
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 73 | 34
percentage of participants | 61.6 | 44.1

13. Secondary Outcome: Percentage Of Participants With A Reduction In Lobular Inflammation At Week 36
Description: The NAS is a histologic scale for NASH activity, which combines into a single score steatosis (Grade 0 to 3), ballooning (Grade 0 to 2), and lobular inflammation (Grade 0 to 3). The endpoint presented the percentage of participants with a reduction in lobular inflammation.
Time Frame: Week 36
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 73 | 34
percentage of participants | 21.9 | 17.6

14. Secondary Outcome: Percentage Of Participants With A Reduction In Hepatocellular Ballooning At Week 36
Description: The NAS is a histologic scale for NASH activity, which combines into a single score steatosis (Grade 0 to 3), ballooning (Grade 0 to 2), and lobular inflammation (Grade 0 to 3). The endpoint presented the percentage of participants with a reduction in hepatocellular ballooning.
Time Frame: Week 36
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 73 | 34
percentage of participants | 58.9 | 58.8

15. Secondary Outcome: Percentage Of Participants Achieving NASH Resolution With At Least 2-Point Reduction In NAS At Week 36
Description: The endpoint presented the percentage of participants achieving NASH resolution with a 2-point reduction at Week 36.
Time Frame: Week 36
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 73 | 34
percentage of participants | 27.4 | 14.7

16. Secondary Outcome: Percent Change From Baseline To Week 12 In High-sensitivity C-reactive Protein (hsCRP)
Description: hsCRP was used as a non-invasive inflammation marker for this study. Blood samples were collected to determine the effect of MGL-3196 on hsCRP.
Time Frame: Week 12
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 79 | 39
percent change | 29.3 (18.36) | 13.2 (25.97)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; LS mean difference in hsCRP between MGL-3196 and placebo at Week 12; Test type: Superiority; p = 0.6155, Linear model; Mean Difference (Net) = 16.0, 95% CI 2-sided [-47.0 to 79.0], Standard Error of Mean 31.81

17. Secondary Outcome: Percent Change From Baseline To Week 36 In hsCRP
Description: as for outcome 16
Time Frame: Week 36
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 79 | 39
percent change | 90.9 (67.52) | 34.0 (96.88)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; LS mean difference in hsCRP between MGL-3196 and placebo at Week 36; Test type: Superiority; p = 0.6311, Linear model; Mean Difference (Net) = 56.9, 95% CI 2-sided [-177.4 to 291.1], Standard Error of Mean 118.09

18. Secondary Outcome: Change From Baseline To Week 12 In Serum Alanine Aminotransferase (ALT)
Description: Blood samples were collected to determine the effect of MGL-3196 on serum ALT.
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: IU/L
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 78 | 38
IU/L | -8.2 (2.7) | -5.2 (3.9)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; LS mean difference in ALT between MGL-3196 and placebo at Week 12; Test type: Superiority; p = 0.5260, Linear model; Mean Difference (Net) = -3.0, 95% CI 2-sided [-12.4 to 6.4], Standard Error of Mean 4.73

19. Secondary Outcome: Change From Baseline To Week 36 In ALT
Description: Blood samples were collected to determine the effect of MGL-3196 on serum ALT.
Time Frame: Week 36
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: IU/L
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 78 | 37
IU/L | -15.4 (4.7) | 11.0 (6.8)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; LS mean difference in ALT between MGL-3196 and placebo at Week 36; Test type: Superiority; p = 0.0019, Linear model; Mean Difference (Net) = -26.4, 95% CI 2-sided [-42.8 to -9.9], Standard Error of Mean 8.29

20. Secondary Outcome: Change From Baseline To Week 12 In Serum Aspartate Aminotransferase (AST)
Description: Blood samples were collected to determine the effect of MGL-3196 on serum AST.
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: IU/L
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 78 | 38
IU/L | -5.8 (1.8) | -1.1 (2.5)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; LS mean difference in AST between MGL-3196 and placebo at Week 12; Test type: Superiority; p = 0.1275, Linear model; Mean Difference (Net) = -4.8, 95% CI 2-sided [-10.9 to 1.4], Standard Error of Mean 3.10

21. Secondary Outcome: Change From Baseline To Week 36 In AST
Description: Blood samples were collected to determine the effect of MGL-3196 on serum AST.
Time Frame: Week 36
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: IU/L
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 78 | 37
IU/L | -7.4 (1.9) | 3.6 (2.8)
Statistical Analysis 1: Comparison: MGL-3196; LS mean difference in ALT between MGL-3196 and placebo at Week 36; Test type: Superiority; p = 0.0016, Linear model; Mean Difference (Net) = -11.1, 95% CI 2-sided [-17.8 to -4.3], Standard Error of Mean 3.42

22. Secondary Outcome: Percent Change From Baseline To Week 12 In Lipid Parameters
Description: Blood samples were collected to determine the effect of MGL-3196 on lipid parameters including low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), non-HDL-C, total cholesterol (TC), triglycerides (TG), apolipoprotein B (ApoB), and Apolipoprotein CIII (ApoCIII).
Time Frame: Week 12
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 79 | 39
percent change
  LDL-C | -10.6 (1.96) | 2.2 (2.79)
  HDL-C | 5.0 (1.91) | 1.8 (2.72)
  non-HDL-C | -12.1 (1.74) | 1.2 (2.47)
  TC | -8.7 (1.37) | 0.9 (1.95)
  TG | -6.8 (4.23) | 9.8 (6.01)
  ApoB | -14.5 (1.59) | 0.8 (2.25)
  ApoCIII | -9.1 (3.23) | 8.7 (4.62)
  Lp(a) | -8.6 (7.54) | 12.3 (10.67)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; LS mean difference in LDL-C between MGL-3196 and placebo at Week 12; Test type: Superiority; p = 0.0002, Linear model; Mean Difference (Net) = -12.9, 95% CI 2-sided [-19.6 to -6.1], Standard Error of Mean 3.41
Statistical Analysis 2: Comparison: MGL-3196 vs Placebo; LS mean difference in HDL-C between MGL-3196 and placebo at Week 12; Test type: Superiority; p = 0.3388, Linear model; Mean Difference (Net) = 3.2, 95% CI 2-sided [-3.4 to 9.8], Standard Error of Mean 3.33
Statistical Analysis 3: Comparison: MGL-3196 vs Placebo; LS mean difference in non-HDL-C between MGL-3196 and placebo at Week 12; Test type: Superiority; p < 0.0001, Linear model; Mean Difference (Net) = -13.4, 95% CI 2-sided [-19.3 to -7.4], Standard Error of Mean 3.02
Statistical Analysis 4: Comparison: MGL-3196 vs Placebo; LS mean difference in TC between MGL-3196 and placebo at Week 12; Test type: Superiority; p = 0.0001, Linear model; Mean Difference (Net) = -9.6, 95% CI 2-sided [-14.3 to -4.9], Standard Error of Mean 2.39
Statistical Analysis 5: Comparison: MGL-3196 vs Placebo; LS mean difference in TG between MGL-3196 and placebo at Week 12; Test type: Superiority; p = 0.0258, Linear model; Mean Difference (Net) = -16.6, 95% CI 2-sided [-31.2 to -2.0], Standard Error of Mean 7.35
Statistical Analysis 6: Comparison: MGL-3196 vs Placebo; LS mean difference in ApoB between MGL-3196 and placebo at Week 12; Test type: Superiority; p < 0.0001, Linear model; Mean Difference (Net) = -15.3, 95% CI 2-sided [-20.8 to -9.9], Standard Error of Mean 2.76
Statistical Analysis 7: Comparison: MGL-3196 vs Placebo; LS mean difference in ApoCIII between MGL-3196 and placebo at Week 12; Test type: Superiority; p = 0.0021, Linear model; Mean Difference (Net) = -17.8, 95% CI 2-sided [-28.9 to -6.6], Standard Error of Mean 5.64
Statistical Analysis 8: Comparison: MGL-3196 vs Placebo; LS mean difference in Lp(a) between MGL-3196 and placebo at Week 12; Test type: Superiority; p = 0.1123, ANOVA; Mean Difference (Net) = -20.9, 95% CI 2-sided [-46.8 to 5.0], Standard Error of Mean 13.06

23. Secondary Outcome: Percent Change From Baseline To Week 36 In Lipid Parameters
Description: Blood samples were collected to determine the effect of MGL-3196 on lipid parameters including LDL-C, HDL-C, non-HDL-C, TC, TG, ApoB, and ApoCIII.
Time Frame: Week 36
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 79 | 39
percent change
  LDL-C | -11.0 (2.14) | 1.5 (3.11)
  HDL-C | 10.5 (3.72) | 12.0 (5.41)
  non-HDL-C | -14.0 (1.90) | 2.1 (2.76)
  TC | -8.9 (1.61) | 3.6 (2.34)
  TG | -19.8 (4.29) | 17.5 (6.24)
  ApoB | -16.5 (1.79) | 0.9 (2.58)
  ApoCIII | -12.0 (3.72) | 24.5 (5.42)
  Lp(a) | 19.0 (10.95) | 39.0 (15.82)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; LS mean difference in LDL-C between MGL-3196 and placebo at Week 36; Test type: Superiority; p = 0.0013, Linear model; Mean Difference (Net) = -12.4, 95% CI 2-sided [-19.9 to -5.0], Standard Error of Mean 3.77
Statistical Analysis 2: Comparison: MGL-3196 vs Placebo; LS mean difference in HDL-C between MGL-3196 and placebo at Week 36; Test type: Superiority; p = 0.8213, Linear model; Mean Difference (Net) = -1.5, 95% CI 2-sided [-14.5 to 11.5], Standard Error of Mean 6.56
Statistical Analysis 3: Comparison: MGL-3196 vs Placebo; LS mean difference in nonHDL-C between MGL-3196 and placebo at Week 36; Test type: Superiority; p < 0.0001, Linear model; Mean Difference (Net) = -16.1, 95% CI 2-sided [-22.7 to -9.4], Standard Error of Mean 3.35
Statistical Analysis 4: Comparison: MGL-3196 vs Placebo; LS mean difference in TC between MGL-3196 and placebo at Week 36; Test type: Superiority; p < 0.0001, Linear model; Mean Difference (Net) = -12.5, 95% CI 2-sided [-18.1 to -6.9], Standard Error of Mean 2.83
Statistical Analysis 5: Comparison: MGL-3196 vs Placebo; LS mean difference in TG between MGL-3196 and placebo at Week 36; Test type: Superiority; p < 0.0001, Linear model; Mean Difference (Net) = -37.3, 95% CI 2-sided [-52.3 to -22.3], Standard Error of Mean 7.58
Statistical Analysis 6: Comparison: MGL-3196 vs Placebo; LS mean difference in ApoB between MGL-3196 and placebo at Week 36; Test type: Superiority; p < 0.0001, Linear model; Mean Difference (Net) = -17.4, 95% CI 2-sided [-23.6 to -11.2], Standard Error of Mean 3.14
Statistical Analysis 7: Comparison: MGL-3196 vs Placebo; LS mean difference in ApoCIII between MGL-3196 and placebo at Week 36; Test type: Superiority; p < 0.0001, Linear model; Mean Difference (Net) = -36.5, 95% CI 2-sided [-49.6 to -23.5], Standard Error of Mean 6.58
Statistical Analysis 8: Comparison: MGL-3196 vs Placebo; LS mean difference in Lp(a) between MGL-3196 and placebo at Week 36; Test type: Superiority; p = 0.3008, ANOVA; Mean Difference (Net) = -20.0, 95% CI 2-sided [-58.2 to 18.2], Standard Error of Mean 19.24

24. Secondary Outcome: Percent Change From Baseline To Week 12 In Lipid Parameter Lipoprotein(a) (Lp[a])
Description: Blood samples were collected to determine the effect of MGL-3196 on lipid parameter Lp(a).
Time Frame: Week 12
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 78 | 39
percent change | -8.6 (7.54) | 12.3 (10.67)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; LS mean difference in Lp(a) between MGL-3196 and placebo at Week 12; Test type: Superiority; p = 0.1123, Linear model; Mean Difference (Net) = -20.9, 95% CI 2-sided [-46.8 to 5.0], Standard Error of Mean 13.06

25. Secondary Outcome: Percent Change From Baseline To Week 36 In Lipid Parameter Lp[a]
Description: Blood samples were collected to determine the effect of MGL-3196 on lipid parameter Lp(a).
Time Frame: Week 36
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 71 | 34
percent change | 19.0 (10.95) | 39.0 (15.82)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; LS mean difference in Lp(a) between MGL-3196 and placebo at Week 36; Test type: Superiority; p = 0.3008, Linear model; Mean Difference (Net) = -20.0, 95% CI 2-sided [-58.2 to 18.2], Standard Error of Mean 19.24

26. Secondary Outcome: Change From Baseline To Week 12 And Week 36 In Cytokeratin-18 (CK-18)
Description: Serum CK-18 fragments, detected using the M30 antibody, is a non-invasive biomarker for NASH that may reflect hepatocyte apoptosis.
Time Frame: Week 12 and Week 36
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 78 | 37
U/L
  Week 12 | -146.2 (35) | -87.5 (51)
  Week 36: number analyzed (Participants) | 75 | 36
  Week 36 | -272.0 (33) | -101.0 (47)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; LS mean difference in CK-18 between MGL-3196 and placebo at Week 12; Test type: Superiority; p = 0.3419, Linear model; Mean Difference (Net) = -58.75, 95% CI 2-sided [-180.70 to 63.21], Standard Error of Mean 61.551
Statistical Analysis 2: Comparison: MGL-3196 vs Placebo; LS mean difference in CK-18 between MGL-3196 and placebo at Week 36; Test type: Superiority; p = 0.0035, Linear model; Mean Difference (Net) = -171.24, 95% CI 2-sided [-285.06 to -57.42], Standard Error of Mean 57.423

27. Secondary Outcome: Change From Baseline To Week 12 And Week 36 In Enhanced Liver Fibrosis (ELF) Test
Description: The ELF Test is a non-invasive blood test that provides a simple, unitless numeric score that is used as a marker of collagen formation and fibrogenic activity and can be used to assess the risk of progression to cirrhosis. Scores below 9.8 indicate low risk of disease progression, and scores above 11.29 indicate high risk. The ELF score is derived from values of three serum biomarkers: hyaluronic acid (HA), procollagen III N-terminal peptide (PIIINP), and tissue inhibitor of metalloproteinase-1 (TIMP-1). The formula is 2.278 + 0.851 × ln(HA) + 0.751 × ln(PIIINP) + 0.394 × ln(TIMP-1); there are no minimum or maximum values.
Time Frame: Week 12 and Week 36
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 40 | 21
score on a scale
  Week 12 | -0.38 (0.09) | -0.02 (0.12)
  Week 36 | -0.66 (0.12) | -0.18 (0.16)
Statistical Analysis 1: Comparison: MGL-3196 vs Placebo; LS mean difference in ELF-test between MGL-3196 and placebo at Week 12; Test type: Superiority; p = 0.0089, Linear model; Mean Difference (Net) = -0.395, 95% CI 2-sided [-0.686 to -0.103], Standard Error of Mean 0.1458
Statistical Analysis 2: Comparison: MGL-3196 vs Placebo; LS mean difference in ELF test between MGL-3196 and placebo at Week 36; Test type: Superiority; p = 0.0174, Linear model; Mean Difference (Net) = -0.484, 95% CI 2-sided [-0.879 to -0.088], Standard Error of Mean 0.1973

28. Secondary Outcome: Change From Baseline To Week 12 And Week 36 In Fibrosis-4 (Fib-4) Score
Description: The Fib-4 score is a scoring system used to estimate the amount of scarring in the liver. It is based on common clinical parameters (age, AST, ALT, and platelets) and has been shown to have the best diagnostic accuracy for advanced fibrosis when compared with other noninvasive clinical scores. Scores are categorized into low (<1.30), indeterminate (1.30-2.67), or high (>2.67) risk of fibrosis. The formula for Fib-4 is: (Age [yr] x AST [U/L]) / ((PLT [109/L]) x (ALT [U/L])½); there are no minimum or maximum values
Time Frame: Week 12 and Week 36
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 79 | 39
score on a scale
  Week 12: number analyzed (Participants) | 77 | 37
  Week 12 | -0.03 (0.386) | 0.05 (0.374)
  Week 36: number analyzed (Participants) | 76 | 36
  Week 36 | 0.02 (0.356) | 0.07 (0.436)

29. Secondary Outcome: Change From Baseline of Thyrotropin at Week 12
Description: Thyrotropin (TSH) was assessed at each study visit.
Time Frame: Baseline up to Week 12
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 78 | 38
mIU/L | 0.096 (0.9136) | -0.101 (0.9742)

30. Secondary Outcome: Change From Baseline of Total Thyroxine at Week 12
Description: Total thyroxine (FT4) was assessed at each study visit.
Time Frame: Baseline up to Week 12
Measure: Mean (Standard Deviation); unit: μg/dL
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 78 | 38
μg/dL | -1.18 (0.958) | -0.07 (0.726)

31. Secondary Outcome: Change From Baseline of Free Thyroxine at Week 12
Description: Free thyroxine (FT4) was assessed at each study visit.
Time Frame: Baseline up to Week 12
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 78 | 38
ng/dL | -0.147 (0.1154) | 0.001 (0.0930)

32. Secondary Outcome: Change From Baseline of Total Triiodothyronine at Week 12
Description: Total Triiodothyronine (T3) was assessed at each study visit.
Time Frame: Baseline up to Week 12
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 78 | 38
μg/L | 0.03 (0.189) | 0.02 (0.236)

33. Secondary Outcome: Change From Baseline of Free Triiodothyronine at Week 12
Description: Free triiodothyronine (T3) was assessed at each study visit.
Time Frame: Baseline up to Week 12
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 78 | 38
ng/L | 0.05 (0.363) | -0.02 (0.513)

34. Secondary Outcome: Change From Baseline of Thyroxine Binding Globulin at Week 12
Description: Thyroxine Binding Globulin was assessed at each study visit.
Time Frame: Baseline up to Week 12
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 78 | 38
mg/L | -1.42 (3.859) | 0.39 (3.522)

35. Secondary Outcome: Change From Baseline of Reverse Triiodothyronine Globulin at Week 12
Description: Reverse Triiodothyronine (T3) was assessed at each study visit.
Time Frame: Baseline up to Week 12
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 78 | 38
ng/dL | -5.22 (5.255) | -0.96 (5.757)

36. Secondary Outcome: Change From Baseline of Thyrotropin at Week 36
Description: Tyrotropin (TSH) was assessed at each study visit.
Time Frame: Baseline up to Week 36
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 79 | 39
mIU/L | 0.034 (0.9705) | 0.043 (0.9481)

37. Secondary Outcome: Change From Baseline of Total Thyroxine at Week 36
Description: Total thyroxine (FT4), thyrotropin (TSH) was assessed at each study visit.
Time Frame: Baseline up to Week 36
Measure: Mean (Standard Deviation); unit: μg/dL
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 79 | 39
μg/dL | -1.10 (1.013) | -0.17 (0.846)

38. Secondary Outcome: Change From Baseline of Free Thyroxine Week 36
Description: Total free thyroxine (FT4) was assessed at each study visit.
Time Frame: Baseline up to Week 36
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 79 | 39
ng/dL | -0.138 (0.1280) | -0.007 (0.1162)

39. Secondary Outcome: Change From Baseline of Total Triiodothyronine at Week 36
Description: Total triiodothyronine (T3) was assessed at each study visit.
Time Frame: Baseline up to Week 36
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 79 | 39
μg/L | 0.02 (0.212) | -0.2 (0.190)

40. Secondary Outcome: Change From Baseline of Free Triiodothyronine at Week 36
Description: Free triiodothyronine (T3) was assessed at each study visit.
Time Frame: Baseline up to Week 36
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 79 | 39
ng/L | 0.02 (0.404) | -0.02 (0.475)

41. Secondary Outcome: Change From Baseline of Thyroxine-Binding Globulin at Week 36
Description: Thyroxine-binding globulin (TBG) was assessed at each study visit.
Time Frame: Baseline up to Week 36
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 79 | 39
mg/L | -0.38 (4.411) | 1.35 (5.639)

42. Secondary Outcome: Change From Baseline of Reverse Triiodothyronine at Week 36
Description: Reverse triiodothyronine (T3) was assessed at each study visit.
Time Frame: Baseline up to Week 36
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | MGL-3196 | Placebo
Number analyzed (Participants) | 79 | 39
ng/dL | -4.41 (5.582) | -1.04 (5.493)

ADVERSE EVENTS:
Time Frame: Screening up to Week 36
Description: Safety population: all randomized participants who received at least 1 dose of study drug. No summaries of AEs by dose level were planned or performed.
Groups:
- MGL-3196 Main Study: Randomized participants received MGL-3196 80 mg orally once daily in the morning for 36 weeks.
- Placebo Main Study: Randomized participants received matching placebo orally once daily in the morning for 36 weeks.
- Extension Study: Patients randomized to MGL-3196 during the Main Study remained on the same dose of MGL-3196 or had a prespecified increase in dose upon entering the Extension Study. Former placebo patients were treated with 80 mg MGL-3196 initially, then up-titrated to 100 mg, remained on 80 mg, or had their dose reduced to 60 mg at Week 4 based on a PK sample obtained during Week 2.
Arm/Group | MGL-3196 Main Study | Placebo Main Study | Extension Study
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/41 | 0/31
Serious Adverse Events (participants affected / at risk) | 5/84 | 2/41 | 0/31
Other Adverse Events (participants affected / at risk) | 73/84 | 28/41 | 6/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MGL-3196 Main Study (N=84) | Placebo Main Study (N=41) | Extension Study (N=31)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bile duct stones (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MGL-3196 Main Study (N=84) | Placebo Main Study (N=41) | Extension Study (N=31)
Diarrhoea (Gastrointestinal disorders) | 31 (49) | 4 (4) | 2 (6)
Nausea (Gastrointestinal disorders) | 17 (17) | 2 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 6 (8) | 3 (3) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 7 (9) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 9 (10) | 4 (6) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 2 (3) | 3 (3)
Influenza (Infections and infestations) | 6 (6) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 11 (14) | 6 (7) | 0 (0)
Dizziness (Nervous system disorders) | 6 (7) | 4 (4) | 0 (0)
Fatigue (General disorders) | 4 (5) | 4 (4) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (6) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release up to 45 days prior to submission and can embargo communications regarding study results for a period that is more than 90 days from the date that the communication is submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot unilaterally extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-12-26): https://cdn.clinicaltrials.gov/large-docs/60/NCT02912260/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT02912260/SAP_001.pdf